CLINICAL TRIAL: NCT00328562
Title: A Phase I Study of ZD1839 (Iressa) and Hypofractionated Thoracic Radiotherapy With Stereotactic Body Frame Immobilization for Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: ZD1839 With Hypofractionated Radiation Therapy With an Immobilization Device for Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03C.225; 2003-07 (Other: CCRRC); JT 1436 (Other: JeffTrial Number)
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Non-Small Cell Lung Carcinoma (NSCLC)
Keywords: Advanced NSCLC; Non-Small Cell Lung Carcinoma; Stage IV NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Iressa and RT (Experimental): Iressa plus thoracic RT at the following dose levels:
  * Level 1: 42.0 Gy in 10 fractions of 4.2 Gy
  * Level 2: 50.4 Gy in 12 fractions of 4.2 Gy
  * Level 3: 63.0 Gy in 15 fractions of 4.2 Gy
  Interventions: Drug: ZD1839 (Iressa); Radiation: Thoracic Radiotherapy

INTERVENTIONS:
Drug: ZD1839 (Iressa)
Radiation: Thoracic Radiotherapy

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of Iressa when used with a short course of high dose radiation therapy in patients with lung cancer.

DETAILED DESCRIPTION:
To estimate treatment-related esophageal, pulmonary, hematologic, and other toxicity of patients with non-small-cell lung cancer (NSCLC) receiving ZD1839 with hypofractionated thoracic radiotherapy (RT). All estimates of toxicity rates will be presented with corresponding confidence intervals using the exact method. The method of Atkinson and Brown will be used due to the two-stage sampling; the method of Conover will be used for tumor response.

To estimate tumor response rates of this treatment regimen and identify the most effective RT dose level, defined as the level associated with the best response rate. Estimates of tumor response rates will be presented with corresponding confidence intervals using the exact method of Conover. Survival will be estimated by the Kaplan-Meier method.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non small cell lung cancer
* Stage IV needing radiation therapy to control symptoms
* Patients with brain metastases
* Unresectable or medically inoperable

Exclusion Criteria:

* Small cell lung cancer
* Previous thoracic radiation therapy
* Oxygen-dependent patients
* Forced expiratory volume in 1 second (FEV1) less than 1.5
* Patients with active interstitial lung disease
* Patients with underlying lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-12; Primary Completion 2008-04 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Werner-Wasik, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University — http://www.kimmelcancercenter.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Iressa and RT
Started | 13
Completed | 12
Not Completed | 1
Not completed — Disease progression | 1

BASELINE CHARACTERISTICS:
Groups:
- Iressa and RT: Iressa plus thoracic RT at the following dose levels:
  * Level 1: 42.0 Gy in 10 fractions of 4.2 Gy
  * Level 2: 50.4 Gy in 12 fractions of 4.2 Gy
  * Level 3: 63.0 Gy in 15 fractions of 4.2 Gy
  ZD1839 (Iressa)
  Thoracic Radiotherapy
Arm/Group | Iressa and RT
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.75 (13.24)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Patients Affected by Treatment-related Morbidities
Description: See "Adverse Events" section for specific toxicities
Time Frame: Twice weekly during RT and at 1-, 2-, 3-, 4-, 5-, and 6-month points after therapy
Measure: Number; unit: participants
Arm/Group | Iressa and RT
Number analyzed (Participants) | 12
participants | 12

2. Secondary Outcome: Tumor Response
Description: Definitions of objective tumor response
  * Complete response - disappearance of all target lesions
  * Partial response - at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter
  * Progressive disease - at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions
  * Stable disease - neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter since the treatment started
Time Frame: Baseline, 1, 3, and 5 months post-treatment
Measure: Number; unit: participants
Arm/Group | Iressa and RT
Number analyzed (Participants) | 12
participants
  Complete response | 3
  Partial response | 1
  Minor response | 3
  Stable disease | 1
  Progressive disease | 1
  Not evaluable | 3

3. Secondary Outcome: Progression-free Survival
Time Frame: Baseline to date of progression
Measure: Median (Full Range); unit: months
Arm/Group | Iressa and RT
Number analyzed (Participants) | 12
months | 5 [2 to 11]

4. Secondary Outcome: Survival From Starting Gefitinib
Time Frame: Baseline to date of expiration
Measure: Median (Full Range); unit: months
Arm/Group | Iressa and RT
Number analyzed (Participants) | 12
months | 10 [1 to 26]

ADVERSE EVENTS:
Arm/Group | Iressa and RT
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iressa and RT (N=12)
Death (General disorders) | 5 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iressa and RT (N=12)
Shoulder pain (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Dysphagia (General disorders) | 4 (4)
Cough (General disorders) | 3 (3)
Nausea (General disorders) | 3 (3)
Diarrhea (General disorders) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Decreased hemoglobin (Blood and lymphatic system disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Increased alkaline phosphatase (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (General disorders) | 1 (1)
Decreased whole blood count (Blood and lymphatic system disorders) | 2 (2)
Weight loss (General disorders) | 2 (2)
Sensory neuropathy (Nervous system disorders) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Side pain (General disorders) | 1 (1)
Bladder pain (General disorders) | 1 (1)
Salivary gland changes (General disorders) | 1 (1)
Alopecia (General disorders) | 1 (1)
Throat pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes